CLINICAL TRIAL: NCT06812351
Title: Clinical and Radiographic Outcome of Regenerative Endodontic Treatment in Immature Permanent Human Teeth Using a Collagen Hydroxyapatite Scaffold
Brief Title: Clinical and Radiographic Outcome of Regeneration in Immature Permanent Human Teeth Using a New Scaffold
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Menna Ali, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT1
Record Dates: First submitted 2024-12-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Randomized Clinical Trial
MeSH Terms: interventions — Blood Coagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaffold with blood clot group (Experimental): root canals were filled with Osteon III Collagen scaffold after blood clot induction during revascularization.
  Interventions: Drug: Osteon III collagen
- blood clot group (Placebo Comparator): root canals were filled with blood clot only after conventional revascularization procedure.
  Interventions: Biological: Blood clot

INTERVENTIONS:
Drug: Osteon III collagen — Hydroxyapatite and tricalcium phosphate particles embeded in bovine collagen
  Other Names: Double antibiotic liquid
  Arms: Scaffold with blood clot group
Biological: Blood clot — Induction of bleeding from apical papilla
  Arms: blood clot group

SUMMARY:
This study aimed to evaluate clinical and radiographic outcome of regeneration in immature permanent human teeth using two different types of scaffolds:

1. Collagen-hydroxyapatite scaffold (Osteon III collagen) after blood clot.
2. Conventional blood clot scaffold.

ELIGIBILITY:
Inclusion Criteria:

1. Single rooted immature permanent teeth.
2. Symptoms:

   1. Pulp necrosis either due to infection or trauma.
   2. Periapical condition; tooth should have periapical radiolucency.
3. Tooth should be restorable without the need for further post placement.
4. Age: from 6-15 years.
5. Sex: males or females.
6. Preoperative Cone beam Computed tomography is a must.

Exclusion Criteria:

* Teeth with complete root formation. 2. Teeth that are badly broken down with difficult isolation. 3. Medically compromised patients. 4. Periodontally affected teeth.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-03-22 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Root completion of immature teeth | 1 year follow up
  Root completion of immature teeth will be measured in terms of increase in root length, dentin thickness and apical foramen closure

SECONDARY OUTCOMES:
positive sensibility test | 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abdelhakim El gendy, PhD, Study Director — AinShams University; Maram Farouk Obeid, PhD, Study Director — AinShams University
Locations (1):
- AinShams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No